CLINICAL TRIAL: NCT01918371
Title: A Retrospective Study of Anti-Vascular Endothelial Growth Factor (VEGF) Injections for Retinal Vein Occlusion or Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-OZU-13-598
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Retinal Vein Occlusion; Macular Edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Bevacizumab; Ranibizumab; aflibercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with RVO: Patients with retinal vein occlusion (RVO) receiving anti-VEGF injection(s) (ranibizumab, bevacizumab or aflibercept) in accordance with standard of care practices. This is a retrospective chart review study.
  Interventions: Drug: Anti-VEGF
- Patients with DME: Patients with diabetic macular edema (DME) receiving anti-VEGF injection(s) (ranibizumab, bevacizumab or aflibercept) in accordance with standard of care practices. This is a retrospective chart review study.
  Interventions: Drug: Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — Patients with retinal vein occlusion or diabetic macular edema receiving anti-VEGF injection(s) in accordance with standard of care practices. This is a retrospective chart review study.
  Other Names: Avastin®; Lucentis®; Eylea®

SUMMARY:
This retrospective data review study will evaluate anti-VEGF injections for retinal vein occlusion (RVO) or diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Macular edema in the study eye due to RVO or DME
* Received an anti-VEGF injection in the study eye on or after June 2010 for RVO and on or after August 2012 for DME

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Received Anti-VEGF injections for retinal vein occlusion (RVO) or diabetic macular edema (DME)
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2014-09-04 (Actual); Study Completion 2014-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Antonio, Texas, United States

REFERENCES:
- [Background] Jumper JM, Dugel PU, Chen S, Blinder KJ, Walt JG. Anti-VEGF treatment of macular edema associated with retinal vein occlusion: patterns of use and effectiveness in clinical practice (ECHO study report 2). Clin Ophthalmol. 2018 Apr 3;12:621-629. doi: 10.2147/OPTH.S163859. eCollection 2018. PMID 29662298

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 323 patients were enrolled in the study and were divided into 2 groups based on their diagnosis: 166 patients with Retinal Vein Occlusion and 157 patients with Diabetic Macular Edema. 2 patients (1 in each group) were missing data and are not included in the analyses.
Period: Overall Study
Arm/Group | Patients With RVO | Patients With DME
Started | 166 | 157
Participants With Complete Data | 165 | 156
Completed | 165 | 156
Not Completed | 1 | 1
Not completed — Missing Data | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants with data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With RVO | Patients With DME | Total
Number analyzed (Participants) | 165 | 156 | 321
Age, Continuous [Mean (Full Range); unit: years] | 69.4 (13.62) [26 to 99] | 63.4 (11.29) [31 to 91] | 66.4 (NA) [26 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 72 | 152
  Male | 85 | 84 | 169

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 2
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). 20/40 or better is equivalent to 14 or more lines read correctly. CRT was measured using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina performed in the study eye after pupil dilation.
Time Frame: Up to Time of Injection 2 (Up to 4 Years)
Population: All participants with data available up to time of Injection 2.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 115 | 104
percentage of participants | 26.09 | 16.35

2. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 3
Description: as for outcome 1
Time Frame: Up to Time of Injection 3 (Up to 4 Years)
Population: All participants with data available up to time of Injection 3.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 118 | 110
percentage of participants | 28.81 | 16.36

3. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 4
Description: as for outcome 1
Time Frame: Up to Time of Injection 4 (Up to 4 Years)
Population: All participants with data available up to time of Injection 4.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 128 | 114
percentage of participants | 26.56 | 17.54

4. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 5
Description: as for outcome 1
Time Frame: Up to Time of Injection 5 (Up to 4 Years)
Population: All participants with data available up to time of Injection 5.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 123 | 95
percentage of participants | 36.59 | 22.11

5. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 6
Description: as for outcome 1
Time Frame: Up to Time of Injection 6 (Up to 4 Years)
Population: All participants with data available up to time of Injection 6.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 106 | 77
percentage of participants | 25.47 | 19.48

6. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 7
Description: as for outcome 1
Time Frame: Up to Time of Injection 7 (Up to 4 Years)
Population: All participants with data available up to time of Injection 7.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 96 | 70
percentage of participants | 32.29 | 20.00

7. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 8
Description: as for outcome 1
Time Frame: Up to Time of Injection 8 (Up to 4 Years)
Population: All participants with data available up to time of Injection 8.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 77 | 48
percentage of participants | 25.97 | 18.75

8. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 9
Description: as for outcome 1
Time Frame: Up to Time of Injection 9 (Up to 4 Years)
Population: All participants with data available up to time of Injection 9.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 64 | 41
percentage of participants | 32.81 | 24.39

9. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 10
Description: as for outcome 1
Time Frame: Up to Time of Injection 10 (Up to 4 Years)
Population: All participants with data available up to time of Injection 10.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 63 | 36
percentage of participants | 28.57 | 22.22

10. Primary Outcome: Percentage of Participants With Best Corrected Visual Acuity (BCVA) of 20/40 or Better and Central Retinal Thickness (CRT) ≤250 µm on Time Domain (TD) Optical Coherence Tomography (OCT) or ≤300 µm on Spectral Domain (SD) OCT Up to Injection 11
Description: as for outcome 1
Time Frame: Up to Time of Injection 11 (Up to 4 Years)
Population: All participants with data available up to time of Injection 11.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 53 | 18
percentage of participants | 28.30 | 38.89

11. Secondary Outcome: Percentage of Participants With BCVA of 20/40 or Better in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). 20/40 or better is equivalent to 14 or more lines read correctly
Time Frame: Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 53.24 | 54.89
  Up to Time of Injection 3 (n=141,135) | 53.19 | 53.33
  Up to Time of Injection 4 (n=141,129) | 50.35 | 51.94
  Up to Time of Injection 5 (n=134,113) | 56.72 | 56.64
  Up to Time of Injection 6 (n=120,101) | 47.50 | 55.45
  Up to Time of Injection 7 (n=107,79) | 48.60 | 54.43
  Up to Time of Injection 8 (n=86,53) | 46.51 | 62.26
  Up to Time of Injection 9 (n=74,45) | 52.70 | 55.56
  Up to Time of Injection 10 (n=65,39) | 43.08 | 53.85
  Up to Time of Injection 11 (n=56,23) | 44.64 | 56.52

12. Secondary Outcome: Percentage of Participants With CRT of ≤250 µm on TD OCT or ≤300 µm on SD OCT in the Study Eye
Description: CRT was measured using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina performed in the study eye after pupil dilation.
Time Frame: Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=133,118) | 50.38 | 28.81
  Up to Time of Injection 3 (n=134,122) | 56.72 | 26.23
  Up to Time of Injection 4 (n=145,129) | 53.10 | 29.46
  Up to Time of Injection 5 (n=137,106) | 59.12 | 33.02
  Up to Time of Injection 6 (n=115,83) | 54.78 | 33.73
  Up to Time of Injection 7 (n=104,80) | 56.73 | 31.25
  Up to Time of Injection 8 (n=85,61) | 57.65 | 27.87
  Up to Time of Injection 9 (n=74,47) | 63.51 | 31.91
  Up to Time of Injection 10(n=74,43) | 67.57 | 27.91
  Up to Time of Injection 11(n=58,25) | 63.79 | 48.0

13. Secondary Outcome: Percentage of Participants With Both BCVA 20/40 or Better or CRT ≤250 µm on TD OCT or ≤300 µm on SD OCT in the Study Eye
Description: as for outcome 1
Time Frame: Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=157,147) | 70.06 | 59.86
  Up to Time of Injection 3 (n=157,147) | 73.25 | 57.82
  Up to Time of Injection 4(n=158,144) | 71.52 | 58.33
  Up to Time of Injection 5 (n=148,124) | 75.68 | 62.10
  Up to Time of Injection 6 (n=129,107) | 71.32 | 63.55
  Up to Time of Injection 7 (n=115,89) | 69.57 | 60.67
  Up to Time of Injection 8 (n=94,66) | 72.34 | 60.61
  Up to Time of Injection 9 (n=84,51) | 77.38 | 58.82
  Up to Time of Injection 10 (n=76,46) | 77.63 | 54.35
  Up to Time of Injection 11 (n=61,30) | 77.05 | 60.00

14. Secondary Outcome: Mean BCVA in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best).
Time Frame: UP to 4 Years
Population: All participants with data available.
Measure: Mean (Standard Deviation); unit: lines
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
lines
  Baseline (n=133,130) | 10.6 (4.04) | 11.8 (3.50)
  Up to Time of Injection 2 (n=139,133) | 12.7 (3.69) | 12.8 (3.38)
  Up to Time of Injection 3 (n=141,135) | 13.0 (3.56) | 12.9 (2.97)
  Up to Time of Injection 4 (n=141,129) | 12.4 (4.09) | 12.9 (3.20)
  Up to Time of Injection 5 (n=134,113) | 12.7 (3.87) | 13.0 (3.02)
  Up to Time of Injection 6 (n=120,101) | 12.5 (3.82) | 12.9 (2.89)
  Up to Time of Injection 7 (n=107,79) | 12.5 (3.97) | 12.8 (3.18)
  Up to Time of Injection 8 (n=86,53) | 12.3 (4.12) | 12.8 (3.37)
  Up to Time of Injection 9 (n=74,45) | 12.7 (3.80) | 12.7 (3.52)
  Up to Time of Injection 10 (n=65,39) | 12.3 (3.49) | 12.3 (3.81)
  Up to Time of Injection 11 (n=56,23) | 12.1 (3.83) | 12.0 (4.88)

15. Secondary Outcome: Change From Baseline in BCVA in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Mean (Standard Deviation); unit: lines
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
lines
  Baseline (n=133,130) | 10.6 (4.04) | 11.8 (3.50)
  Change from Baseline Up to Injection 2(n=116,114) | 1.6 (3.12) | 1.0 (2.46)
  Change from Baseline Up to Injection 3 (n=115,117) | 1.9 (3.33) | 1.3 (2.63)
  Change from Baseline Up to Injection 4 (n=118,109) | 1.6 (3.37) | 1.1 (2.51)
  Change from Baseline Up to Injection 5 (n=109,98) | 1.7 (4.02) | 1.3 (2.62)
  Change from Baseline Up to Injection 6 (n=101,86) | 1.9 (4.18) | 1.2 (2.48)
  Change from Baseline Up to Injection 7 (n=89,69) | 2.1 (4.04) | 1.1 (2.31)
  Change from Baseline Up to Injection 8 (n=73,43) | 1.7 (4.32) | 0.8 (2.65)
  Change from Baseline Up to Injection 9 (n=66,37) | 1.9 (4.00) | 1.5 (3.19)
  Change from Baseline Up to Injection 10 (n=58,33) | 1.8 (3.96) | 1.3 (3.46)
  Change from Baseline Up to Injection 11 (n=49,17) | 1.4 (4.21) | 0.4 (3.73)

16. Secondary Outcome: Percentage of Participants With an Increase From Baseline of ≥2 Lines in BCVA in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). An increase of 2 or more lines read correctly from Baseline indicates improvement.
Time Frame: Baseline, Up to 4 Years
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 40.29 | 30.08
  Up to Time of Injection 3 (n=141,135) | 40.43 | 35.56
  Up to Time of Injection 4 (n=141,129) | 40.43 | 29.46
  Up to Time of Injection 5 (n=134,113) | 40.30 | 32.74
  Up to Time of Injection 6 (n=120,101) | 40.83 | 25.74
  Up to Time of Injection 7 (n=107,79) | 46.73 | 35.44
  Up to Time of Injection 8 (n=86,53) | 46.51 | 28.30
  Up to Time of Injection 9 (n=74,45) | 50.00 | 33.33
  Up to Time of Injection 10 (n=65,39) | 47.69 | 33.33
  Up to Time of Injection 11 (n=56,23) | 41.07 | 21.74

17. Secondary Outcome: Percentage of Participants With an Increase From Baseline of ≥3 Lines in BCVA in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). An increase of 3 or more lines read correctly from Baseline indicates improvement.
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 25.90 | 14.29
  Up to Time of Injection 3 (n=141,135) | 28.37 | 20.00
  Up to Time of Injection 4 (n=141,129) | 25.53 | 17.83
  Up to Time of Injection 5 (n=134,113) | 32.09 | 20.35
  Up to Time of Injection 6 (n=120,101) | 30.83 | 19.80
  Up to Time of Injection 7 (n=107,79) | 36.45 | 21.52
  Up to Time of Injection 8 (n=86,53) | 30.23 | 22.64
  Up to Time of Injection 9 (n=74,45) | 40.54 | 28.89
  Up to Time of Injection 10 (n=65,39) | 40.00 | 28.21
  Up to Time of Injection 11 (n=56,23) | 35.71 | 17.39

18. Secondary Outcome: Change From Baseline in CRT by OCT in the Study Eye
Description: CRT was measured using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina performed in the study eye after pupil dilation. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Mean (Standard Deviation); unit: µm (microns)
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
µm (microns)
  Baseline (n=128,119) | 499.1 (188.14) | 413.4 (104.85)
  Change from Baseline Up to Injection 2 (n=110,95) | -159.5 (183.98) | -44.7 (93.62)
  Change from Baseline Up to Injection 3 (n=110,95) | -158.6 (188.06) | -62.1 (100.61)
  Change from Baseline Up to Injection4 (n=117,104) | -151.9 (204.10) | -66.8 (102.31)
  Change from Baseline Up to Injection 5 (n=109,84) | -169.4 (211.28) | -55.7 (82.23)
  Change from Baseline Up to Injection 6 (n=93,68) | -180.8 (223.14) | -63.0 (89.54)
  Change from Baseline Up to Injection 7 (n=85,67) | -171.5 (225.49) | -70.1 (97.13)
  Change from Baseline Up to Injection 8 (n=70,47) | -202.7 (191.62) | -82.5 (103.79)
  Change from Baseline Up to Injection 9 (n=63,37) | -224.2 (186.64) | -66.4 (108.21)
  Change from Baseline Up to Injection 10 (n=65,31) | -210.0 (226.05) | -60.9 (105.07)
  Change from Baseline Up to Injection 11 (n=48,18) | -212.4 (207.39) | -76.0 (119.54)

19. Secondary Outcome: Time to Improvement of ≥2 Lines in BCVA in the Study Eye
Description: Kaplan-Meier estimates of the time in months to improvement of ≥2 lines in BCVA. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best).
Time Frame: 4 Years
Population: All participants with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months | 4.6667 [0.0000 to 44.6333] | 7.1500 [0.0000 to 45.033]

20. Secondary Outcome: Time to Improvement of ≥3 Lines in BCVA in the Study Eye
Description: Kaplan-Meier estimates of the time in months to improvement of ≥3 lines in BCVA. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best).
Time Frame: 4 Years
Population: All participants with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months | 7.2167 [0.0000 to 44.6333] | 9.1000 [0.233 to 843.700]

21. Secondary Outcome: Time to Improvement in BCVA to 20/40 or Better in the Study Eye
Description: Kaplan-Meier estimates of the time to Improvement in months in BCVA to 20/40 or Better. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). 20/40 or better is equivalent to 14 or more lines read correctly.
Time Frame: 4 Years
Population: All participants with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months | 2.3167 [0.0667 to 44.6333] | 3.3667 [0.000 to 843.700]

22. Secondary Outcome: Time to Improvement in CRT of ≤250 µm on TD OCT or ≤300 µm on SD OCT in the Study Eye
Description: Kaplan-Meier estimates of the time to improvement in months in CRT of ≤250 µm on TD OCT or ≤300 µm on SD OCT. CRT was measured using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina performed in the study eye after pupil dilation.
Time Frame: 4 Years
Population: All participants with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months | 2.5333 [0.2333 to 45.7333] | 7.9333 [0.233 to 854.133]

23. Secondary Outcome: Time to Improvement to Both 20/40 or Better in BCVA and Improvement in CRT of ≤250 µm on TD OCT or ≤300 µm on SD OCT in the Study Eye
Description: Kaplan-Meier estimates of the time to improvement to Both 20/40 or Better in BCVA and Improvement in CRT of ≤250 µm on TD OCT or ≤300 µm on SD OCT. BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). 20/40 or better is equivalent to 14 or more lines read correctly. CRT was measured using OCT, a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina performed in the study eye after pupil dilation.
Time Frame: 4 Years
Population: All participants with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months | 7.6167 [0.2333 to 45.7333] | 9.8000 [0.233 to 854.133]

24. Secondary Outcome: Time Between Anti-VEGF Injections in the Study Eye
Description: The mean time in months between anti-VEGF Injections.
Time Frame: 4 Years
Population: All participants with data available.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
months
  Up to Time of Injection 2 (n=163,152) | 1.1 (0.57) | 1.5 (1.38)
  Up to Time of Injection 3 (n=162,154) | 1.1 (0.60) | 1.6 (1.32)
  Up to Time of Injection 4 (n=157,141) | 1.4 (1.10) | 1.7 (1.49)
  Up to Time of Injection 5 (n=143,124) | 1.3 (0.73) | 1.4 (0.97)
  Up to Time of Injection 6 (n=127,106) | 1.4 (1.19) | 1.3 (0.60)
  Up to Time of Injection 7 (n=114,89) | 1.5 (1.70) | 1.5 (1.20)
  Up to Time of Injection 8 (n=99,64) | 1.6 (3.11) | 1.3 (0.59)
  Up to Time of Injection 9 (n=82,52) | 1.3 (0.78) | 1.4 (1.12)
  Up to Time of Injection 10 (n=73,40) | 1.4 (0.57) | 1.2 (0.64)
  Up to Time of Injection 11 (n=63,30) | 1.3 (0.53) | 1.2 (0.80)

25. Secondary Outcome: Number of Intravitreal Anti-VEGF Injections in the Study Eye
Description: To be included in the time period analysis, patients must have been enrolled on the study for at least a minimum of 0 weeks, 24 weeks, 50 weeks, 100 weeks, and 150 weeks, respectively, and must have received at least 1 injection during that time period.
Time Frame: 0-6 Months, 7-12 Months, Years 1,2,3
Population: All participants with data available.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
injections
  0-6 Months (n = 158,149) | 4.4 (1.40) | 4.0 (1.64)
  7-12 Months (n = 99,64) | 3.3 (1.64) | 2.8 (1.42)
  Year 1 (n = 117,80) | 7.1 (2.90) | 5.8 (2.77)
  Year 2 (n = 40,23) | 5.4 (2.98) | 5.0 (2.65)
  Year 3 (n = 17,10) | 5.9 (2.99) | 3.4 (1.96)

26. Secondary Outcome: Percentage of Participants Switching to a Second or Third Anti-VEGF Agent After First Injection in the Study Eye
Time Frame: UP to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 155
percentage of participants | 33.33 | 47.44

27. Secondary Outcome: Percentage of Participants Switching Among Different Anti-VEGF Agents in the Study Eye
Description: Participants who switched among the different Anti-VEGF Agents: bevacizumab, ranibizumab and aflibercept.
Time Frame: Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  bevacizumab to aflibercept | 2.67 | 0.0
  bevacizumab to ranibizumab | 13.33 | 25.26
  aflibercept to bevacizumab | 4.00 | 0.0
  aflibercept to ranibizumab | 20.00 | 1.05
  ranibizumab to bevacizumab | 53.33 | 73.68
  ranibizumab to aflibercept | 6.67 | 0.0

28. Secondary Outcome: Percentage of Participants Undergoing Focal Laser Surgery in the Study Eye
Time Frame: 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants | 20.00 | 44.87

29. Secondary Outcome: Percentage of Participants Undergoing Panretinal Photocoagulation (PRP) Surgery in the Study Eye
Time Frame: 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants | 5.45 | 13.46

30. Secondary Outcome: Percentage of Participants With a Loss (Decrease) in BCVA of ≥1 Line From Baseline in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). A loss of 1 or more lines read correctly from Baseline indicates a worsening of vision.
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 13.67 | 15.79
  Up to Time of Injection 3 (n=141,135) | 14.18 | 21.48
  Up to Time of Injection 4 (n=141,129) | 20.57 | 23.26
  Up to Time of Injection 5 (n=134,113) | 20.15 | 15.04
  Up to Time of Injection 6 (n=120,101) | 17.50 | 19.80
  Up to Time of Injection 7 (n=107,79) | 18.69 | 18.99
  Up to Time of Injection 8 (n=86,53) | 16.28 | 22.64
  Up to Time of Injection 9 (n=74,45) | 14.86 | 17.78
  Up to Time of Injection 10 (n=65,39) | 21.54 | 20.51
  Up to Time of Injection 11 (n=56,23) | 23.21 | 13.04

31. Secondary Outcome: Percentage of Participants With a Gain (Increase) in BCVA of ≥1 Line From Baseline in the Study Eye
Description: BCVA was assessed using the Snellen eye chart converted to Early Treatment Diabetic Retinopathy Study number of lines ranging from 0 (worst) to 20 (best). A gain of 1 or more lines read correctly from Baseline indicates an improvement of vision.
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 58.99 | 45.86
  Up to Time of Injection 3 (n=141,135) | 61.70 | 53.33
  Up to Time of Injection 4 (n=141,129) | 55.32 | 47.29
  Up to Time of Injection 5 (n=134,113) | 53.73 | 50.44
  Up to Time of Injection 6 (n=120,101) | 55.83 | 44.55
  Up to Time of Injection 7 (n=107,79) | 58.88 | 45.57
  Up to Time of Injection 8 (n=86,53) | 54.65 | 45.28
  Up to Time of Injection 9 (n=74,45) | 59.46 | 44.44
  Up to Time of Injection 10 (n=65,39) | 60.00 | 41.03
  Up to Time of Injection 11 (n=56,23) | 55.36 | 39.13

32. Secondary Outcome: Percentage of Participants With No Change in BCVA From Baseline in the Study Eye
Description: as for outcome 14
Time Frame: Baseline, Up to 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants
  Up to Time of Injection 2 (n=139,133) | 17.99 | 34.59
  Up to Time of Injection 3 (n=141,135) | 14.89 | 19.26
  Up to Time of Injection 4 (n=141,129) | 16.31 | 25.58
  Up to Time of Injection 5 (n=134,113) | 17.16 | 24.78
  Up to Time of Injection 6 (n=120,101) | 16.67 | 23.76
  Up to Time of Injection 7 (n=107,79) | 12.15 | 30.38
  Up to Time of Injection 8 (n=86,53) | 18.60 | 18.87
  Up to Time of Injection 9 (n=74,45) | 18.92 | 31.11
  Up to Time of Injection 10 (n=65,39) | 13.85 | 30.77
  Up to Time of Injection 11 (n=56,23) | 16.07 | 21.74

33. Secondary Outcome: Percentage of Participants Undergoing Glaucoma Laser Surgery in the Study Eye
Time Frame: 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants | 0.61 | 0.64

34. Secondary Outcome: Percentage of Participants Undergoing Incisional Glaucoma Surgery in the Study Eye
Time Frame: 4 Years
Population: All participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 165 | 156
percentage of participants | 1.21 | 0.00

35. Secondary Outcome: Percentage of Phakic Patients With Cataract Surgery in the Study Eye
Description: Phakic patients have intraocular lens implants.
Time Frame: 4 Years
Population: All phakic participants with data available.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With RVO | Patients With DME
Number analyzed (Participants) | 117 | 104
percentage of participants | 17.0 | 15.0

ADVERSE EVENTS:
Time Frame: Up to 4 Years
Arm/Group | Patients With RVO | Patients With DME
Serious Adverse Events (participants affected / at risk) | 12/165 | 12/156
Other Adverse Events (participants affected / at risk) | 0/165 | 0/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With RVO (N=165) | Patients With DME (N=156)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Hospitalized for sepsis (Infections and infestations) | 0 | 1
Pacemaker placed (Surgical and medical procedures) | 0 | 1
Patient was hospitalized for dizziness (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Soft tissue mass cancer right leg (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 1 | 2
Unknown heart complications (Cardiac disorders) | 0 | 2
Bowel obstruction (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fluid in lungs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hositalized for heart problems (Cardiac disorders) | 1 | 0
Hospitalized for lack of oxygen (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperallergic reaction to iron (Immune system disorders) | 1 | 0
Methicilin-resistant staphylococcus aureus (Infections and infestations) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Retinal detachment OS (left eye) (Eye disorders) | 1 | 0
Spots of blurred vision in left eye (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.